CLINICAL TRIAL: NCT05291520
Title: A Phase 1, Open-Label, Single-Dose Study of the Safety and Pharmacokinetics of a Human Monoclonal Antibody, GSK3810109, Administered Either Subcutaneously or Intravenously With Recombinant Human Hyaluronidase PH20 (rHuPH20) to Healthy Adults
Brief Title: A Study to Investigate the Safety and Pharmacokinetics of a Single Dose of VH3810109 (Also Known as GSK3810109), Administered Either Subcutaneously (SC) With rHuPH20 or Intravenously (IV), in Healthy Adult Participants
Acronym: SPAN
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 217901
Record Dates: First submitted 2022-02-16; First posted 2022-03-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: HIV Infections
Keywords: VH3810109; GSK3810109; HIV; Human Monoclonal Antibody; rHuPH20; Pharmacokinetics; Safety; Tolerability; N6LS
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Intervention Model Description: Participants will receive a single SC or IV dose of VH3810109 co-administered with rHuPH20
Masking Description: This will be an open-label study. Hence, there will be no masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] (Experimental): Participants in this group received a single subcutaneous (SC) dose of VH3810109 20 mg/kg co-administered with rHuPH20 at Day 1 and were followed up to 24 weeks.
  Interventions: Biological: VH3810109; Biological: rHuPH20
- Part 2 Group: VH3810109 60 mg/kg [IV] (Experimental): Participants in this group received a single intravenous (IV) dose of VH3810109 60 mg/kg at Day 1 and were followed up to 24 weeks.
  Interventions: Biological: VH3810109
- Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC] (Experimental): Participants in this group received a single subcutaneous (SC) dose of VH3810109 3000 mg co-administered with rHuPH20 at Day 1 and were followed up to 24 weeks.
  Interventions: Biological: VH3810109; Biological: rHuPH20

INTERVENTIONS:
Biological: VH3810109 — VH3810109 was administered.
Biological: rHuPH20 — rHuPH20 was administered.
  Arms: Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC]; Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]

SUMMARY:
An open-label, two part study to assess the safety, tolerability, and PK of VH3810109 in healthy adult participants. Participants will receive a single SC or IV dose of VH3810109 co-administered with rHuPH20 and will be followed up for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and without history of any of the conditions listed in the exclusion criteria.
* Participants having body weight of ≥50 kilogram (kg) and <100 kg
* Participants having a clinical laboratory profile within the normal range or must have results that do not show clinically significant abnormalities, as judged by the investigator at screening.
* Contraceptive use by men or women participants should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

Participants who are female at birth are eligible to participate if at least one of the following conditions applies:

Not pregnant or breastfeeding and at least one of the following conditions applies:

Is not a participant of childbearing potential (POCBP) or Is a POCBP and agree to use an acceptable contraceptive method as described in Section 10.4 from 3 weeks prior to the start of this study and during the study. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

A POCBP must have a negative highly sensitive serum pregnancy test on Day -1, prior to the first dose of study intervention All participants in the study should be counseled on safer sexual practices including the use and benefit/risk of effective barrier methods (e.g., male condom).

The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a POCBP with an early undetected pregnancy.

* Capable of giving written informed consent.

Exclusion Criteria:

* Hypertension that is not well controlled.
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, hematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study intervention or interfering with the interpretation of data.
* Positive human immunodeficiency virus (HIV) antibody test.
* Positive test result for SARS-CoV-2.
* Evidence of hepatitis B (HB) virus infection at screening or within 3 months prior to first dose of study intervention Participants positive for Hepatitis B antigen (HBsAg) are excluded. Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status) and positive for Hepatitis B virus (HBV) DNA are excluded
* Any history of a severe allergic reaction with generalized urticaria, angioedema or anaphylaxis within the 2 years prior to enrollment that has a reasonable risk of recurrence during the study.
* The participant has an underlying skin disease or disorder (i.e., infection, inflammation, dermatitis, eczema, drug rash, drug allergy, psoriasis, food allergy, urticaria) or tattoos that would interfere with assessment of injection sites.
* History of sensitivity to any of the study medications or their components or drugs of their class, or a history of drug or other allergy that, in the opinion of the investigator or medical monitor, contraindicates their participation.
* Clinically significant multiple or severe drug allergies, intolerance to topical corticosteroids, or severe post-treatment hypersensitivity reactions (including, but not limited to, erythema multiforme major, linear immunoglobulin A, dermatosis, toxic epidermal necrolysis, and exfoliative dermatitis).
* Exposure to an experimental drug, human blood product, or vaccine (which does not have emergency, conditional, or standard market authorization) within 28 days prior to the first dose of study treatment OR plans to receive live vaccines during the study.
* Prior receipt of licensed or investigational Monoclonal antibody (Mab).
* Receipt of any investigational study agent within 28 days prior to first dose of study treatment
* Prior exposure to VH3810109 or rHuPH20 in this or another clinical study.
* Where participation in the study would result in donation of blood or blood products in excess of 500 milliliter (mL) within 56 days.
* Exposure to more than 4 new chemical entities within 12 months prior to the first dosing day.
* ALT ≥1.5 times the upper limit of normal (ULN).
* Total bilirubin ≥1.5 times the ULN (isolated total bilirubin >1.5×ULN is acceptable if total bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Corrected QT interval Fridericia's formula (QTcF)>450 millisecond (msec) for males and QTcF >470 msec for females.
* The participant has a tattoo or other dermatological condition overlying potential injection sites that may interfere with interpretation of ISRs or administration of VH3810109.
* Grade 4 laboratory abnormalities.
* Any other chronic or clinically significant medical condition that in the opinion of investigator would jeopardize the safety or rights of the subject including (but not limited to): diabetes mellitus type I, chronic hepatitis; OR clinically significant forms of drug or alcohol abuse, asthma, autoimmune disease, psychiatric disorders, heart disease, or cancer.
* Known hypersensitivity to hyaluronidase or any of the excipients in ENHANZ Drug Product (EDP)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — ViiV Healthcare
Locations (1):
- GSK Investigational Site, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Leone PA, Losos J, Wannamaker P, D'Agostino R, Warwick-Sanders M, Ghita GL, Wilches V, Donatti C, Brown K, Gandhi Y. VH3810109 (N6LS) broadly neutralizing antibody safety, pharmacokinetics, and anti-drug antibody incidence in adults without HIV: phase 1 SPAN study results. Antimicrob Agents Chemother. 2025 Sep 3;69(9):e0025825. doi: 10.1128/aac.00258-25. Epub 2025 Jul 23. PMID 40698814

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Started | 8 | 8 | 8
Completed | 8 | 8 | 7
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC] | Total
Number analyzed (Participants) | 8 | 8 | 8 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.8 (7.76) | 40.0 (14.45) | 39.9 (10.59) | 40.87 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 3 | 15
  Male | 3 | 1 | 5 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 2 | 1 | 1 | 4
  Black or African American | 1 | 2 | 4 | 7
  White | 5 | 4 | 3 | 12
  Multiple | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Grade 2 or Higher (>=) Adverse Events (AEs) Following SC Administration of VH3810109 (Part 1 and Part 3)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. The Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric AE was used for all AE severity grading, where Grade 1=Mild, 2=Moderate, 3=Severe, 4=Potentially life threatening. This outcome measure is presenting only data for Grade 2 or more of severity.
Time Frame: Up to Week 24
Population: Analysis was performed on the Safety set which included all participants that received at least one dose of the study intervention and had data for the assessed timepoints and analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Participants | 7 | 8

2. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) Following SC Administration of VH3810109 (Part 1 and Part 3)
Description: An SAE is defined as any untoward medical occurrence that; results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect or other situations as judged by physician.
Time Frame: Up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Injection Site Reactions (ISRs) Following VH3810109 SC Administration (Part 1 and 3)
Description: ISRs were recorded via ISR diaries and managed through investigator assessment. The participants who experienced any injection site reaction were reported.
Time Frame: Up to 7 days post-dose
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Participants | 7 | 8

4. Primary Outcome: Number of Participants With Grade 2 to 4 Elevated Alanin Aminotransferase/Aspartate Aminotransferase (ALT/AST) Values Following VH3810109 SC Administration (Part 1 and 3)
Description: Liver chemistry stopping and increased monitoring criteria is analyzed using DAIDS AE Grading Table, where Grade 2 (moderate): causing greater than minimal interference with usual social and functional activities, Grade 3 (severe): causing inability to perform usual social and functional activities, Grade 4 (Potentially life threatening): causing inability to perform basic self-care functions or hospitalization indicated.
Time Frame: Up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Participants
  ALT, Grade 2 | 0 | 0
  ALT, Grade 3 | 0 | 0
  ALT, Grade 4 | 0 | 0
  AST, Grade 2 | 0 | 0
  AST, Grade 3 | 0 | 0
  AST, Grade 4 | 0 | 0

5. Primary Outcome: Number of Participants With >= Grade 2 AEs Following IV Administration of VH3810109 (Part 2)
Description: as for outcome 1
Time Frame: Up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Group: VH3810109 60 mg/kg [IV]
Number analyzed (Participants) | 8
Participants | 0

6. Primary Outcome: Number of Participants With SAEs Following IV Administration of VH3810109 (Part 2)
Description: as for outcome 2
Time Frame: Up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Group: VH3810109 60 mg/kg [IV]
Number analyzed (Participants) | 8
Participants | 0

7. Primary Outcome: Number of Participants With Grade 2 to 4 Elevated ALT/AST Values Following VH3810109 IV Administration (Part 2)
Description: as for outcome 4
Time Frame: Up to Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2 Group: VH3810109 60 mg/kg [IV]
Number analyzed (Participants) | 8
Participants
  ALT, Grade 2 | 0
  ALT, Grade 3 | 0
  ALT, Grade 4 | 0
  AST, Grade 2 | 0
  AST, Grade 3 | 0
  AST, Grade 4 | 0

8. Secondary Outcome: Area Under the Plasma Concentration-time Curve (AUC) From Time Zero Extrapolated to Infinity (AUC[0-inf]) of VH3810109
Description: Blood samples were collected as assessed by protocol, at specific time points for pharmacokinetic (PK) analysis of VH3810109.
Time Frame: Up to Week 24
Population: Analysis was performed on PK Parameter Analysis Set, which included participants who received study intervention and for whom valid and evaluable serum PK parameters were derived for the assessed timepoints and analysis.
Measure: Mean (95% Confidence Interval); unit: Day*microgram/mililitre (day*μg/mL)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Day*microgram/mililitre (day*μg/mL) | 7587 [4789 to 10380] | 31560 [27620 to 35490] | 12840 [8883 to 16800]

9. Secondary Outcome: AUC From Time Zero to Time t (AUC[0-t]) of VH3810109
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis of VH3810109.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: day*μg/mL
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
day*μg/mL | 6996 [4512 to 9479] | 29160 [25550 to 32770] | 11590 [7819 to 15360]

10. Secondary Outcome: Maximum Observed Concentration (Cmax) of VH3810109
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis of VH3810109.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
μg/mL | 148.2 [117.3 to 179.1] | 1864 [1620 to 2107] | 321.1 [201.6 to 440.6]

11. Secondary Outcome: Time of Maximum Observed Concentration (Tmax) of VH3810109
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis of VH3810109.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Days | 4.503 [1.472 to 7.535] | 0.046 [0.045 to 0.047] | 2.882 [2.586 to 3.178]

12. Secondary Outcome: Apparent Terminal Phase Half-life (t1/2) of VH3810109
Description: Blood samples were collected as assessed by protocol, at specific time points for PK analysis of VH3810109.
Time Frame: Up to Week 24
Population: as for outcome 8
Measure: Mean (95% Confidence Interval); unit: Days
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Days | 38.17 [23.41 to 52.93] | 46.97 [40.86 to 53.09] | 44.95 [34.14 to 55.76]

13. Secondary Outcome: Score Recorded for "Acceptance of ISRs", Using Perception of Injection (PIN) Questionnaire (Part 1 and 3)
Description: The PIN questionnaire measure contains 21 items: pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside clinical trial. Scores range from 1 to 5; questions are phrased to ensure that 1: most favorable perception of vaccination, and 5: most unfavorable. Score of a dimension is calculated as mean of all items with dimension. Higher scores represent worse perception of injection.
Time Frame: At Day 2 and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Scores on a scale
  Acceptance of ISRs, Day 2 | 1.44 (1.050) | 1.44 (0.496)
  Acceptance of ISRs, Day 7 | 1.44 (0.729) | 1.50 (0.802)

14. Secondary Outcome: Number of Participants Reporting Pain, Using Perception of Injection (PIN) Questionnaire (Part 1 and 3)
Description: The PIN questionnaire measure contains 21 items: pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside clinical trial.
  Scores range from 1 to 5; the scores are defined as following: 1=not at all bothered, 2=a little bothered, 3=moderately bothered, 4=very bothered, 5=extremely bothered; questions are phrased to ensure that 1: most favorable perception of vaccination, and 5: most unfavorable. Score of a dimension is calculated as mean of all items with dimension. Higher scores represent worse perception of injection.
Time Frame: At Day 2 and Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Participants
  Not at all bothered by pain, Day 2 | 6 | 6
  A little bothered by pain, Day 2 | 2 | 2
  Moderately bothered by pain, Day 2 | 0 | 0
  Very bothered by pain, Day 2 | 0 | 0
  Extremely bothered by pain, Day 2 | 0 | 0
  Not at all bothered by pain, Day 7 | 5 | 5
  A little bothered by pain, Day 7 | 3 | 3
  Moderately bothered by pain, Day 7 | 0 | 0
  Very bothered by pain, Day 7 | 0 | 0
  Extremely bothered by pain, Day 7 | 0 | 0

15. Secondary Outcome: Number of Participants Reporting Being Bothered or Affected by the Pain and Local Reactions Based on the PIN Questionaire (Part 1 and 3)
Description: The PIN questionnaire measure contains 21 items: pain at injection site, local site reactions, impact on functioning and willingness to pursue injectable treatment outside clinical trial.
  Scores range from 1 to 5; the scores are defind as following: 1=totaly acceptable, 2=very acceptable, 3=moderately acceptable, 4=a little acceptable, 5=not at all acceptable; questions are phrased to ensure that 1: most favorable perception of vaccination, and 5: most unfavorable. Score of a dimension is calculated as mean of all items with dimension. Higher scores represent worse perception of injection.
Time Frame: At Day 2 and Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Participants
  Totally acceptable local reactions, Day 2 | 7 | 6
  Very acceptable local reactions, Day 2 | 0 | 1
  Moderately acceptable local reactions, Day 2 | 0 | 1
  A little acceptable local reactions, Day 2 | 1 | 0
  Not at all acceptable local reactions, Day 2 | 0 | 0
  Totally acceptable local reactions, Day 7 | 5 | 6
  Very acceptable local reactions, Day 7 | 2 | 1
  Moderately acceptable local reactions, Day 7 | 1 | 1
  A little acceptable local reactions, Day 7 | 0 | 0
  Not at all acceptable local reactions, Day 7 | 0 | 0
  Totally acceptable pain, Day 2 | 6 | 4
  Very acceptable pain, Day 2 | 1 | 4
  Moderately acceptable pain, Day 2 | 0 | 0
  A little acceptable pain, Day 2 | 1 | 0
  Not at all acceptable pain, Day 2 | 0 | 0
  Totally acceptable pain, Day 7 | 6 | 5
  Very acceptable pain, Day 7 | 1 | 1
  Moderately acceptable pain, Day 7 | 1 | 2
  A little acceptable pain, Day 7 | 0 | 0
  Not at all acceptable pain, Day 7 | 0 | 0

16. Secondary Outcome: Score Reported for Post-injection Pain Assessment Using Numeric Rating Scale (NRS) Following VH3810109 SC Administration (Part 1 and 3)
Description: Post-injection assessment of pain was measured based on NRS which is a 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst possible pain).
Time Frame: At Day 1, Day 2 and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Scores on a scale
  Day 1 | 3.63 (2.326) | 2.75 (2.550)
  Day 2 | 3.63 (2.615) | 0.63 (0.744)
  Day 7 | 3.63 (2.925) | 0.38 (0.744)

17. Secondary Outcome: Scores Reported for Post-injection Pain Assessment Using Numeric Rating Scale (NRS) Following VH3810109 IV Administration (Part 2)
Description: as for outcome 16
Time Frame: At Day 1, Day 2 and Day 7
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Part 2 Group: VH3810109 60 mg/kg [IV]
Number analyzed (Participants) | 8
Scores on a scale
  Day 1 | 0.50 (1.069)
  Day 2 | 0.88 (1.642)
  Day 7 | 0.50 (1.414)

18. Secondary Outcome: Number of ISRs Events Overall and by Grade (Part 1 and 3)
Description: ISRs were recorded via ISR diaries and managed through investigator assessment. Severity of injection site reactions was analyzed using DAIDS AE Grading Table. The severity was categorized into grades as following: Grade 1 (mild): causing no or minimal interference with usual social and functional activities, Grade 2 (moderate): causing greater than minimal interference with usual social and functional activities, Grade 3 (severe): causing inability to perform usual social and functional activities, Grade 4 (Potentially life threatening): causing inability to perform basic self-care functions or hospitalization indicated, Grade 5 (death). Higher grade indicates more severe condition.
Time Frame: Up to day 14
Population: as for outcome 1
Measure: Count of Units; unit: Number of events
Units Other Than Participants: Number of events
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Number analyzed (Number of events) | 14 | 18
Number of events
  Overall ISRs | 14 | 18
  Grade 1 ISRs | 2 | 6
  Grade 2 ISRs | 5 | 2
  Grade 3 ISRs | 7 | 10
  Grade 4 ISRs | 0 | 0
  Grade 5 ISRs | 0 | 0

19. Secondary Outcome: The Overall Duration of ISRs, Expressed in Days
Description: ISRs will be recorded via ISR diaries and managed through investigator assessment.
Time Frame: From Day 1 up to Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8
Days | 2.9 (1.35) | 4.6 (6.29)

20. Secondary Outcome: Change From Baseline in Platelets, White Blood Cells (WBC), Neutrophils, Lymphocytes, Monocytes, Eosinophils and Basophils
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: Analysis was performed on PK set, who included participants who received study intervention and for whom valid and evaluable serum PK parameters were derived for the assesseed timepoints and analysis.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
10^9 cells/L
  Basophils, at Baseline | 0.033 (0.0139) | 0.035 (0.0207) | 0.044 (0.0106)
  Basophils, at Day 2 | -0.004 (0.0092) | 0.000 (0.0151) | -0.009 (0.0083)
  Basophils, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Basophils, at Day 3 |  | 0.005 (0.0152) | -0.009 (0.0113)
  Basophils, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Basophils, at Day 4 |  | 0.012 (0.0172) | -0.001 (0.0181)
  Basophils, at Day 7 | 0.008 (0.0128) | 0.003 (0.0128) | -0.005 (0.0107)
  Basophils, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Basophils, at Day 8 |  | 0.002 (0.0098) |
  Basophils, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Basophils, at Day 10 |  | 0.000 (0.0283) |
  Basophils, at Day 14 | 0.001 (0.0064) | 0.008 (0.0139) | 0.003 (0.0149)
  Basophils, at Week 4 | 0.003 (0.0139) | 0.004 (0.0141) | 0.000 (0.0185)
  Basophils, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Basophils, at Week 16 | -0.001 (0.0083) | 0.004 (0.0192) | -0.001 (0.0121)
  Basophils, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Basophils, at Week 24 | 0.000 (0.0151) | 0.001 (0.0259) | -0.013 (0.0160)
  Eosinophils, at Baseline | 0.121 (0.0957) | 0.098 (0.0333) | 0.145 (0.1370)
  Eosinophils, at Day 2 | 0.018 (0.0851) | 0.010 (0.0151) | 0.016 (0.0385)
  Eosinophils, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Eosinophils, at Day 3 |  | 0.017 (0.0121) | 0.010 (0.0513)
  Eosinophils, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Eosinophils, at Day 4 |  | 0.022 (0.0194) | 0.010 (0.0431)
  Eosinophils, at Day 7 | 0.016 (0.0964) | 0.000 (0.0293) | 0.016 (0.0619)
  Eosinophils, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Eosinophils, at Day 8 |  | 0.003 (0.0320) |
  Eosinophils, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Eosinophils, at Day 10 |  | -0.010 (0.0424) |
  Eosinophils, at Day 14 | 0.059 (0.0718) | 0.011 (0.0624) | 0.025 (0.0444)
  Eosinophils, at Week 4 | 0.045 (0.0644) | 0.001 (0.0290) | -0.004 (0.0403)
  Eosinophils, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Eosinophils, at Week 16 | 0.059 (0.1667) | 0.053 (0.1269) | 0.013 (0.0605)
  Eosinophils, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Eosinophils, at Week 24 | 0.001 (0.1063) | 0.094 (0.1445) | -0.001 (0.0527)
  WBC, at Baseline | 5.13 (1.161) | 6.31 (1.365) | 6.50 (2.036)
  WBC, at Day 2 | 0.43 (0.696) | -0.31 (1.253) | -0.36 (0.980)
  WBC, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  WBC, at Day 3 |  | 0.13 (1.113) | -0.41 (1.089)
  WBC, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  WBC, at Day 4 |  | 0.32 (1.386) | -0.49 (1.360)
  WBC, at Day 7 | 0.11 (0.872) | -0.04 (1.171) | -0.25 (2.165)
  WBC, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  WBC, at Day 8 |  | -0.05 (0.997) |
  WBC, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  WBC, at Day 10 |  | -0.85 (0.071) |
  WBC, at Day 14 | -0.26 (0.809) | -0.38 (0.791) | -0.25 (0.994)
  WBC, at Week 4 | -0.03 (1.261) | -0.40 (0.857) | -0.48 (1.340)
  WBC, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  WBC, at Week 16 | 0.01 (0.892) | -0.63 (1.073) | -0.64 (1.162)
  WBC, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  WBC, at Week 24 | -0.46 (0.883) | 0.40 (2.438) | -0.51 (0.540)
  Lymphocytes, at Baseline | 1.368 (0.2680) | 2.214 (0.5545) | 2.086 (0.4824)
  Lymphocytes, at Day 2 | 0.006 (0.1908) | -0.484 (0.3503) | -0.094 (0.2147)
  Lymphocytes, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Lymphocytes, at Day 3 |  | -0.175 (0.3459) | -0.135 (0.2727)
  Lymphocytes, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Lymphocytes, at Day 4 |  | -0.065 (0.3551) | -0.106 (0.3847)
  Lymphocytes, at Day 7 | -0.043 (0.1763) | -0.211 (0.3189) | -0.175 (0.3166)
  Lymphocytes, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Lymphocytes, at Day 8 |  | -0.193 (0.3462) |
  Lymphocytes, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Lymphocytes, at Day 10 |  | -0.475 (0.0778) |
  Lymphocytes, at Day 14 | -0.019 (0.1664) | -0.386 (0.3366) | -0.161 (0.3561)
  Lymphocytes, at Week 4 | 0.063 (0.1943) | -0.314 (0.2911) | -0.226 (0.2908)
  Lymphocytes, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Lymphocytes, at Week 16 | 0.100 (0.2441) | -0.190 (0.2478) | -0.191 (0.3559)
  Lymphocytes, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Lymphocytes, at Week 24 | 0.058 (0.3377) | -0.380 (0.3497) | -0.339 (0.4461)
  Monocytes, at Baseline | 0.396 (0.1556) | 0.461 (0.1038) | 0.485 (0.1488)
  Monocytes, at Day 2 | 0.091 (0.1037) | -0.048 (0.1159) | -0.008 (0.0587)
  Monocytes, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Monocytes, at Day 3 |  | 0.040 (0.0639) | -0.013 (0.0886)
  Monocytes, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Monocytes, at Day 4 |  | 0.080 (0.0957) | -0.006 (0.1034)
  Monocytes, at Day 7 | 0.049 (0.1185) | -0.021 (0.1572) | -0.013 (0.1413)
  Monocytes, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Monocytes, at Day 8 |  | 0.008 (0.1019) |
  Monocytes, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Monocytes, at Day 10 |  | -0.110 (0.1131) |
  Monocytes, at Day 14 | 0.034 (0.1347) | -0.078 (0.1237) | -0.015 (0.1319)
  Monocytes, at Week 4 | 0.036 (0.1061) | -0.045 (0.1146) | -0.034 (0.1010)
  Monocytes, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Monocytes, at Week 16 | 0.023 (0.0630) | -0.029 (0.1221) | 0.001 (0.0724)
  Monocytes, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Monocytes, at Week 24 | -0.018 (0.1099) | 0.001 (0.1670) | -0.020 (0.0462)
  Neutrophils, at Baseline | 3.218 (0.9157) | 3.499 (0.9783) | 3.756 (1.6757)
  Neutrophils, at Day 2 | 0.315 (0.8333) | 0.214 (1.0869) | -0.263 (0.9093)
  Neutrophils, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Neutrophils, at Day 3 |  | 0.238 (0.9621) | -0.291 (0.9503)
  Neutrophils, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Neutrophils, at Day 4 |  | 0.262 (1.0730) | -0.398 (1.0114)
  Neutrophils, at Day 7 | 0.066 (0.8177) | 0.210 (0.9063) | -0.079 (1.8480)
  Neutrophils, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Neutrophils, at Day 8 |  | 0.160 (0.8802) |
  Neutrophils, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Neutrophils, at Day 10 |  | -0.270 (0.3111) |
  Neutrophils, at Day 14 | -0.340 (0.7531) | 0.096 (0.8912) | -0.116 (0.7571)
  Neutrophils, at Week 4 | -0.160 (1.2887) | -0.036 (0.9269) | -0.233 (1.1531)
  Neutrophils, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Neutrophils, at Week 16 | -0.178 (0.6481) | -0.468 (0.9437) | -0.500 (0.9401)
  Neutrophils, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Neutrophils, at Week 24 | -0.535 (0.8511) | 0.691 (2.3541) | -0.160 (0.6340)
  Platelets, at Baseline | 256.3 (48.96) | 301.9 (34.84) | 289.5 (71.95)
  Platelets, at Day 2 | 6.6 (12.70) | -14.6 (12.95) | 1.0 (18.48)
  Platelets, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Platelets, at Day 3 |  | 3.2 (19.77) | 0.1 (19.63)
  Platelets, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Platelets, at Day 4 |  | -4.2 (17.22) | -4.9 (20.16)
  Platelets, at Day 7 | 1.4 (13.65) | 0.0 (13.49) | 1.9 (23.46)
  Platelets, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Platelets, at Day 8 |  | 2.8 (12.14) |
  Platelets, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Platelets, at Day 10 |  | -8.0 (19.80) |
  Platelets, at Day 14 | 19.9 (32.89) | 1.0 (52.60) | 2.1 (40.86)
  Platelets, at Week 4 | 30.6 (87.1) | -3.5 (15.10) | 3.1 (31.31)
  Platelets, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Platelets, at Week 16 | -0.5 (19.34) | 6.6 (35.49) | -6.4 (31.43)
  Platelets, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Platelets, at Week 24 | 1.1 (27.58) | 12.5 (37.14) | -2.3 (27.79)

21. Secondary Outcome: Change From Baseline in Hematocrit
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: Analysis was performed on PK set, who included participants who received study intervention and for whom valid and evaluable serum PK parameters were derived for the assessed timepoints and analysis.
Measure: Mean (Standard Deviation); unit: Proportion of red blood cells in blood
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Proportion of red blood cells in blood
  Baseline | 0.3873 (0.04541) | 0.3928 (0.04415) | 0.4253 (0.04709)
  Day 2 | 0.0159 (0.02226) | 0.0005 (0.01513) | 0.0118 (0.01704)
  Day 3: number analyzed (Participants) | 0 | 6 | 8
  Day 3 |  | 0.0100 (0.02612) | 0.0066 (0.01502)
  Day 4: number analyzed (Participants) | 0 | 6 | 8
  Day 4 |  | 0.0003 (0.01992) | 0.0023 (0.01646)
  Day 7 | 0.0168 (0.01662) | 0.0043 (0.01521) | -0.0065 (0.01208)
  Day 8: number analyzed (Participants) | 0 | 6 | 0
  Day 8 |  | 0.0062 (0.01781) |
  Day 10: number analyzed (Participants) | 0 | 2 | 0
  Day 10 |  | -0.0270 (0.01131) |
  Day 14 | 0.0118 (0.01426) | -0.0074 (0.01736) | -0.0056 (0.01420)
  Week 4 | 0.0016 (0.01672) | -0.0013 (0.01641) | -0.0069 (0.01605)
  Week 16: number analyzed (Participants) | 8 | 8 | 7
  Week 16 | 0.0196 (0.02303) | 0.0078 (0.02315) | -0.0106 (0.00759)
  Week 24: number analyzed (Participants) | 8 | 8 | 7
  Week 24 | 0.0119 (0.01389) | 0.0053 (0.02437) | -0.0076 (0.03243)

22. Secondary Outcome: Change From Baseline in Hemoglobin, Albumin and Total Protein
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Grams per liter (g/L)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Grams per liter (g/L)
  Hemoglobin, at Baseline | 131.4 (16.78) | 128.3 (15.83) | 142.4 (15.67)
  Hemoglobin, at Day 2 | 5.8 (6.90) | 1.9 (4.61) | 3.9 (6.49)
  Hemoglobin, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Hemoglobin, at Day 3 |  | 6.8 (6.79) | 4.3 (5.39)
  Hemoglobin, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Hemoglobin, at Day 4 |  | 4.8 (7.19) | 3.9 (5.46)
  Hemoglobin, at Day 7 | 2.6 (6.35) | 2.9 (5.28) | -0.4 (4.37)
  Hemoglobin, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Hemoglobin, at Day 8 |  | 3.3 (4.84) |
  Hemoglobin, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Hemoglobin, at Day 10 |  | -10.0 (4.24) |
  Hemoglobin, at Day 14 | 3.4 (4.78) | -0.8 (5.90) | -0.4 (4.47)
  Hemoglobin, at Week 4 | 1.0 (5.29) | 0.4 (6.55) | -1.4 (4.96)
  Hemoglobin, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Hemoglobin, at Week 16 | 4.3 (7.23) | 5.3 (8.01) | -3.4 (4.12)
  Hemoglobin, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Hemoglobin, at Week 24 | 0.4 (4.07) | 4.0 (7.54) | -1.4 (13.99)
  Albumin, at Baseline | 44.0 (3.02) | 43.9 (3.00) | 43.9 (3.44)
  Albumin, at Day 2 | 0.4 (2.07) | -2.4 (2.45) | -0.3 (1.83)
  Albumin, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Albumin, at Day 3 |  | -0.3 (1.86) | -0.1 (1.73)
  Albumin, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Albumin, at Day 4 |  | -0.8 (2.40) | 0.3 (1.58)
  Albumin, at Day 7 | 0.1 (2.80) | -1.9 (1.81) | 0.4 (2.00)
  Albumin, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Albumin, at Day 8 |  | -1.7 (1.75) |
  Albumin, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Albumin, at Day 10 |  | -5.5 (0.71) |
  Albumin, at Day 14 | 0.0 (2.00) | -1.0 (1.51) | -0.1 (1.89)
  Albumin, at Week 4 | -1.4 (2.56) | -0.1 (2.10) | -0.3 (2.43)
  Albumin, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Albumin, at Week 16 | 0.6 (1.77) | 0.8 (2.19) | -2.0 (2.16)
  Albumin, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Albumin, at Week 24 | -1.5 (2.14) | -0.3 (1.04) | -1.9 (2.48)
  Total Protein, at Baseline | 70.0 (3.85) | 71.0 (3.66) | 72.3 (4.40)
  Total Protein, at Day 2 | 0.6 (4.17) | -1.4 (4.17) | -1.5 (3.51)
  Total Protein, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Total Protein, at Day 3 |  | 1.3 (3.93) | -1.9 (3.04)
  Total Protein, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Total Protein, at Day 4 |  | 0.0 (4.43) | 0.6 (2.20)
  Total Protein, at Day 7 | 0.0 (4.57) | -2.8 (2.76) | -0.1 (3.52)
  Total Protein, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Total Protein, at Day 8 |  | 2.76 (2.86) |
  Total Protein, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Total Protein, at Day 10 |  | -8.0 (0.00) |
  Total Protein, at Day 14 | 0.0 (4.14) | -1.6 (2.56) | -0.8 (2.71)
  Total Protein, at Week 4 | -0.6 (3.16) | -1.0 (3.38) | -1.9 (3.14)
  Total Protein, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Total Protein, at Week 16 | 0.9 (2.42) | 1.0 (3.85) | -4.4 (3.87)
  Total Protein, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Total Protein, at Week 24 | -3.4 (3.96) | 0.1 (2.17) | -2.7 (4.46)

23. Secondary Outcome: Change From Baseline in Red Blood Cell Count (RBC)
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Trillion cells/L (TI/L)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Trillion cells/L (TI/L)
  Baseline | 4.518 (0.5518) | 4.523 (0.4014) | 4.889 (0.6362)
  Day 2 | 0.180 (0.2654) | 0.043 (0.1717) | 0.141 (0.2154)
  Day 3: number analyzed (Participants) | 0 | 6 | 8
  Day 3 |  | 0.163 (0.3064) | 0.079 (0.1890)
  Day 4: number analyzed (Participants) | 0 | 6 | 8
  Day 4 |  | 0.085 (0.2239) | 0.056 (0.2169)
  Day 7 | 0.155 (0.2067) | 0.084 (0.1584) | -0.074 (0.1429)
  Day 8: number analyzed (Participants) | 0 | 6 | 0
  Day 8 |  | 0.088 (0.1877) |
  Day 10: number analyzed (Participants) | 0 | 2 | 0
  Day 10 |  | -0.315 (0.1626) |
  Day 14 | 0.130 (0.1646) | -0.088 (0.1940) | -0.064 (0.1686)
  Week 4 | 0.050 (0.1802) | -0.026 (0.1625) | -0.078 (0.1814)
  Week 16: number analyzed (Participants) | 8 | 8 | 7
  Week 16 | 0.186 (0.2612) | 0.124 (0.2212) | -0.164 (0.0752)
  Week 24: number analyzed (Participants) | 8 | 8 | 7
  Week 24 | 0.063 (0.1496) | 0.078 (0.2326) | -0.110 (0.3089)

24. Secondary Outcome: Change From Baseline in Mean Corpuscle Volume (MCV)
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: cubic microns
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
cubic microns
  Baseline | 85.78 (2.013) | 86.89 (6.081) | 87.28 (3.478)
  Day 2 | 0.14 (0.466) | -0.66 (0.478) | -0.03 (0.354)
  Day 3: number analyzed (Participants) | 0 | 6 | 8
  Day 3 |  | -0.72 (0.492) | -0.03 (0.345)
  Day 4: number analyzed (Participants) | 0 | 6 | 8
  Day 4 |  | -1.38 (0.542) | -0.41 (0.589)
  Day 7 | 0.84 (0.661) | -0.61 (0.562) | -0.10 (0.469)
  Day 8: number analyzed (Participants) | 0 | 6 | 0
  Day 8 |  | -0.27 (0.674) |
  Day 10: number analyzed (Participants) | 0 | 2 | 0
  Day 10 |  | 0.05 (0.354) |
  Day 14 | 0.06 (0.784) | 0.04 (0.746) | 0.06 (0.623)
  Week 4 | -0.53 (1.216) | 0.34 (1.125) | -0.03 (0.703)
  Week 16: number analyzed (Participants) | 8 | 8 | 7
  Week 16 | 0.76 (0.842) | -0.75 (2.522) | 0.74 (1.078)
  Week 24: number analyzed (Participants) | 8 | 8 | 7
  Week 24 | 1.34 (1.983) | -0.41 (2.107) | 0.40 (2.195)

25. Secondary Outcome: Change From Baseline in Mean Corpuscle Hemoglobin (MCH)
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: picograms (pg)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
picograms (pg)
  Baseline | 29.05 (1.028) | 28.33 (2.213) | 29.26 (1.660)
  Day 2 | 0.20 (0.553) | 0.21 (0.458) | -0.08 (0.345)
  Day 3: number analyzed (Participants) | 0 | 6 | 8
  Day 3 |  | 0.63 (0.836) | 0.39 (0.290)
  Day 4: number analyzed (Participants) | 0 | 6 | 8
  Day 4 |  | 0.67 (0.463) | 0.55 (0.678)
  Day 7 | -0.36 (0.302) | 0.16 (0.385) | 0.29 (0.536)
  Day 8: number analyzed (Participants) | 0 | 6 | 0
  Day 8 |  | 0.27 (0.480) |
  Day 10: number analyzed (Participants) | 0 | 2 | 0
  Day 10 |  | -0.20 (0.141) |
  Day 14 | -0.06 (0.475) | 0.44 (0.524) | 0.33 (0.590)
  Week 4 | -0.09 (0.608) | 0.39 (0.617) | 0.16 (0.466)
  Week 16: number analyzed (Participants) | 8 | 8 | 7
  Week 16 | -0.21 (0.613) | 0.39 (0.779) | 0.24 (0.737)
  Week 24: number analyzed (Participants) | 8 | 8 | 7
  Week 24 | -0.39 (1.051) | 0.39 (0.716) | 0.31 (1.524)

26. Secondary Outcome: Change From Baseline in Glucose (Fasting), Blood Urea Nitrogen (BUN), Creatinine, Direct Bilirubin and Total Bilirubin
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: milligram per deciliter (mg/dL)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
milligram per deciliter (mg/dL)
  Glucose, at Baseline | 5.009778 (0.2649736) | 5.037533 (0.2582430) | 4.864064 (0.2032812)
  Glucose, at Day 2 | -0.006939 (0.2306696) | 0.256734 (0.5881647) | 0.145714 (0.2966207)
  Glucose, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Glucose, at Day 3 |  | -0.018503 (0.2930311) | 0.201224 (0.3645321)
  Glucose, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Glucose, at Day 4 |  | -0.027755 (0.2868315) | -0.006939 (0.2852734)
  Glucose, at Day 7 | 0.180408 (0.1723749) | 0.548161 (1.1531574) | 0.166530 (0.3408978)
  Glucose, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Glucose, at Day 8 |  | -0.111020 (0.3330600) |
  Glucose, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Glucose, at Day 10 |  | 0.000000 (0.1570060) |
  Glucose, at Day 14 | -0.027755 (0.2586688) | 0.048571 (0.3884992) | 0.006939 (0.2790329)
  Glucose, at Week 4 | 0.027755 (0.3857275) | -0.124898 (0.2842106) | 0.215101 (0.5168587)
  Glucose, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Glucose, at Week 16 | -0.180408 (0.2254827) | 0.076326 (0.2138345) | 0.111020 (0.3376541)
  Glucose, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Glucose, at Week 24 | -0.249795 (0.3040408) | -0.208163 (0.3557469) | 0.237900 (0.3184202)
  Blood urea nitrogen, at Baseline | 3.83775 (0.731134) | 4.19475 (1.376981) | 4.73025 (1.594955)
  Blood urea nitrogen, at Day 2 | 1.21380 (0.678703) | 0.39270 (0.937762) | 0.27221 (1.307383)
  Blood urea nitrogen, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Blood urea nitrogen, at Day 3 |  | 0.67830 (0.651268) | 0.16511 (1.369415)
  Blood urea nitrogen, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Blood urea nitrogen, at Day 4 |  | 0.82705 (0.927490) | 0.15619 (1.726718)
  Blood urea nitrogen, at Day 7 | 0.30345 (1.042747) | 0.58459 (1.250583) | -0.42840 (1.421995)
  Blood urea nitrogen, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Blood urea nitrogen, at Day 8 |  | 0.55930 (0.809900) |
  Blood urea nitrogen, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Blood urea nitrogen, at Day 10 |  | 0.35700 (0.000000) |
  Blood urea nitrogen, at Day 14 | 0.02678 (0.714446) | -0.33915 (1.192768) | -0.50873 (1.656633)
  Blood urea nitrogen, at Week 4 | 0.31684 (0.895135) | -0.16065 (0.695659) | -0.24098 (1.082288)
  Blood urea nitrogen, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Blood urea nitrogen, at Week 16 | 0.21420 (1.260309) | -0.41948 (0.805711) | 0.03060 (1.359639)
  Blood urea nitrogen, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Blood urea nitrogen, at Week 24 | 0.32576 (1.074638) | 0.26775 (1.474420) | -0.05610 (1.187055)
  Creatinine, at Baseline | 68.2890 (15.18504) | 68.0680 (13.56381) | 73.8140 (15.20157)
  Creatinine, at Day 2 | 1.4365 (8.05969) | -3.2045 (3.97975) | 2.3205 (9.02667)
  Creatinine, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Creatinine, at Day 3 |  | -0.7367 (6.16058) | 3.6465 (5.49905)
  Creatinine, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Creatinine, at Day 4 |  | -0.5893 (6.03887) | 0.8840 (7.94898)
  Creatinine, at Day 7 | 0.0000 (5.84472) | 2.4310 (6.71158) | 6.2985 (9.30077)
  Creatinine, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Creatinine, at Day 8 |  | -0.4420 (6.01510) |
  Creatinine, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Creatinine, at Day 10 |  | 11.9340 (3.12541) |
  Creatinine, at Day 14 | 0.1105 (3.82236) | 0.6630 (6.49175) | 3.4255 (5.98510)
  Creatinine, at Week 4 | 2.9835 (7.05521) | 0.1105 (4.18485) | 2.7625 (6.78911)
  Creatinine, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Creatinine, at Week 16 | -0.3315 (6.87895) | -0.7735 (7.98314) | 3.1571 (5.32501)
  Creatinine, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Creatinine, at Week 24 | 2.0995 (4.25102) | -0.2210 (5.62574) | 5.6829 (7.60201)
  Direct Bilirubin, at Baseline | 2.0306 (0.49592) | 1.7741 (0.62621) | 2.1161 (1.04191)
  Direct Bilirubin, at Day 2 | -0.5771 (0.42811) | -0.2138 (0.45473) | -0.0214 (0.44250)
  Direct Bilirubin, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Direct Bilirubin, at Day 3 |  | -0.1425 (0.45134) | -0.1069 (0.43776)
  Direct Bilirubin, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Direct Bilirubin, at Day 4 |  | 0.0285 (0.47656) | 0.1283 (0.58348)
  Direct Bilirubin, at Day 7 | 0.0000 (0.43836) | 0.0214 (0.42320) | -0.1283 (0.33893)
  Direct Bilirubin, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Direct Bilirubin, at Day 8 |  | 0.1995 (0.53440) |
  Direct Bilirubin, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Direct Bilirubin, at Day 10 |  | -0.5130 (0.48366) |
  Direct Bilirubin, at Day 14 | -0.2351 (0.57763) | -0.3634 (0.46997) | -0.1710 (0.44778)
  Direct Bilirubin, at Week 4 | -0.5344 (0.62287) | 0.0000 (0.42872) | -0.1496 (0.50427)
  Direct Bilirubin, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Direct Bilirubin, at Week 16 | -0.3206 (0.59544) | -0.2138 (0.52308) | -0.7817 (0.56591)
  Direct Bilirubin, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Direct Bilirubin, at Week 24 | -0.3420 (0.49222) | -0.2565 (0.61993) | -0.3176 (0.36178)
  Total bilirubin, at Baseline | 9.7684 (3.95623) | 10.4738 (3.28512) | 12.5258 (7.47987)
  Total bilirubin, at Day 2 | -1.9879 (2.22382) | -1.1115 (3.08613) | 0.6413 (2.98813)
  Total bilirubin, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Total bilirubin, at Day 3 |  | -0.8550 (2.99128) | 0.4061 (3.48526)
  Total bilirubin, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Total bilirubin, at Day 4 |  | 0.0570 (2.84018) | 2.0306 (4.64850)
  Total bilirubin, at Day 7 | 1.6031 (2.82603) | -0.2565 (3.16102) | -0.4703 (2.08181)
  Total bilirubin, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Total bilirubin, at Day 8 |  | 0.9405 (3.54057) |
  Total bilirubin, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Total bilirubin, at Day 10 |  | -2.3085 (1.81373) |
  Total bilirubin, at Day 14 | 0.6199 (3.02728) | -2.4368 (2.07377) | -0.6199 (3.52222)
  Total bilirubin, at Week 4 | -1.7528 (3.77392) | -1.1115 (1.51851) | -0.3206 (3.67145)
  Total bilirubin, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Total bilirubin, at Week 16 | -0.4061 (3.45758) | -1.5390 (2.90772) | -2.4917 (2.46196)
  Total bilirubin, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Total bilirubin, at Week 24 | 0.0428 (2.98813) | -0.6840 (3.10368) | -1.6856 (2.63700)

27. Secondary Outcome: Change From Baseline in Sodium, Potassium, Calcium, Chloride and Carbon Dioxide
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Millimole per liter (mmol/L)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Millimole per liter (mmol/L)
  Calcium, at Baseline | 2.329706 (0.1049575) | 2.317231 (0.0805028) | 2.351538 (0.0931159)
  Calcium, at Day 2 | -0.015594 (0.1041067) | -0.003119 (0.0983979) | -0.003119 (0.0983979)
  Calcium, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Calcium, at Day 3 |  | 0.037425 (0.1101762) | 0.003119 (0.0759557)
  Calcium, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Calcium, at Day 4 |  | 0.008317 (0.1145166) | 0.040544 (0.0729700)
  Calcium, at Day 7 | -0.012475 (0.0533453) | -0.006238 (0.0830180) | 0.037425 (0.0442316)
  Calcium, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Calcium, at Day 8 |  | -0.004158 (0.0639356) |
  Calcium, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Calcium, at Day 10 |  | -0.112275 (0.0882116) |
  Calcium, at Day 14 | 0.009356 (0.0398698) | -0.034306 (0.0923367) | -0.009356 (0.0923367)
  Calcium, at Week 4 | -0.031188 (0.0739536) | -0.034306 (0.0853291) | 0.003119 (0.0826826)
  Calcium, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Calcium, at Week 16 | -0.015594 (0.0842805) | 0.018713 (0.0751464) | -0.064157 (0.0496021)
  Calcium, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Calcium, at Week 24 | -0.056138 (0.0861717) | -0.031188 (0.0371268) | -0.053464 (0.1002445)
  Carbon Dioxide, at Baseline | 29.4 (1.77) | 27.8 (2.25) | 28.6 (1.92)
  Carbon Dioxide, at Day 2 | 0.5 (1.41) | 0.6 (1.19) | 0.4 (1.41)
  Carbon Dioxide, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Carbon Dioxide, at Day 3 |  | 1.5 (0.84) | -0.5 (0.93)
  Carbon Dioxide, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Carbon Dioxide, at Day 4 |  | 1.3 (1.03) | 0.3 (1.28)
  Carbon Dioxide, at Day 7 | -0.3 (1.39) | 0.3 (1.28) | 0.3 (0.71)
  Carbon Dioxide, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Carbon Dioxide, at Day 8 |  | 1.3 (1.03) |
  Carbon Dioxide, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Carbon Dioxide, at Day 10 |  | 0.0 (1.41) |
  Carbon Dioxide, at Day 14 | 0.3 (0.89) | 0.5 (1.51) | -0.4 (1.41)
  Carbon Dioxide, at Week 4 | 1.5 (1.51) | 0.9 (1.64) | 0.0 (0.93)
  Carbon Dioxide, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Carbon Dioxide, at Week 16 | -1.3 (1.28) | 0.3 (0.71) | -0.4 (0.98)
  Carbon Dioxide, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Carbon Dioxide, at Week 24 | -0.5 (1.20) | 0.4 (1.51) | 0.3 (1.38)
  Chloride, at Baseline | 103.1 (1.81) | 102.1 (2.59) | 102.4 (2.20)
  Chloride, at Day 2 | -0.6 (2.45) | 0.0 (2.00) | 0.1 (2.42)
  Chloride, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Chloride, at Day 3 |  | -1.2 (1.94) | -0.3 (2.49)
  Chloride, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Chloride, at Day 4 |  | -1.5 (1.64) | -0.4 (2.39)
  Chloride, at Day 7 | -0.5 (1.07) | 0.1 (1.64) | 0.5 (2.14)
  Chloride, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Chloride, at Day 8 |  | 0.3 (1.75) |
  Chloride, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Chloride, at Day 10 |  | 5.5 (2.12) |
  Chloride, at Day 14 | -1.6 (1.77) | 1.0 (2.56) | 0.4 (2.13)
  Chloride, at Week 4 | -1.3 (2.38) | 1.1 (2.47) | 0.4 (1.06)
  Chloride, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Chloride, at Week 16 | -0.4 (2.13) | 1.5 (1.41) | 0.7 (1.80)
  Chloride, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Chloride, at Week 24 | -0.1 (2.36) | 0.6 (2.26) | 1.7 (2.21)
  Potassium, at Baseline | 4.36 (0.484) | 4.14 (0.342) | 4.29 (0.485)
  Potassium, at Day 2 | 0.09 (0.242) | 0.16 (0.325) | 0.10 (0.366)
  Potassium, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Potassium, at Day 3 |  | 0.13 (0.372) | 0.14 (0.250)
  Potassium, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Potassium, at Day 4 |  | 0.00 (0.544) | 0.13 (0.320)
  Potassium, at Day 7 | -0.30 (0.421) | 0.29 (0.470) | -0.01 (0.340)
  Potassium, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Potassium, at Day 8 |  | 0.07 (0.207) |
  Potassium, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Potassium, at Day 10 |  | 0.45 (0.354) |
  Potassium, at Day 14 | -0.13 (0.381) | 0.04 (0.513) | 0.09 (0.458)
  Potassium, at Week 4 | -0.16 (0.389) | 0.18 (0.183) | -0.01 (0.196)
  Potassium, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Potassium, at Week 16 | -0.38 (0.413) | 0.11 (0.189) | -0.04 (0.382)
  Potassium, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Potassium, at Week 24 | -0.06 (0.245) | -0.03 (0.354) | 0.01 (0.308)
  Sodium, at Baseline | 138.8 (1.39) | 137.1 (2.23) | 136.9 (2.53)
  Sodium, at Day 2 | -0.4 (2.13) | -0.4 (2.26) | 0.1 (2.30)
  Sodium, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  Sodium, at Day 3 |  | -0.8 (0.98) | -0.3 (1.49)
  Sodium, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  Sodium, at Day 4 |  | -1.3 (2.25) | -0.1 (1.89)
  Sodium, at Day 7 | -0.5 (1.77) | 0.5 (2.20) | 0.8 (1.98)
  Sodium, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  Sodium, at Day 8 |  | 0.3 (1.51) |
  Sodium, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Sodium, at Day 10 |  | 4.5 (4.95) |
  Sodium, at Day 14 | -1.3 (1.39) | 1.0 (2.88) | 0.6 (1.85)
  Sodium, at Week 4 | -0.9 (2.17) | 1.0 (2.45) | 0.9 (1.64)
  Sodium, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Sodium, at Week 16 | -0.8 (1.58) | 1.0 (2.51) | 1.3 (1.60)
  Sodium, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Sodium, at Week 24 | -1.1 (2.53) | 0.1 (3.48) | 2.0 (2.24)

28. Secondary Outcome: Change From Baseline in ALT, AST and Alkaline Phosphatase (ALP)
Description: Blood samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: International Units per liter (IU/L)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
International Units per liter (IU/L)
  ALT, at Baseline | 11.8 (2.71) | 12.5 (4.00) | 20.0 (8.09)
  ALT, at Day 2 | 0.6 (1.69) | -0.5 (1.31) | -1.8 (3.45)
  ALT, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  ALT, at Day 3 |  | 0.5 (1.52) | -1.1 (4.61)
  ALT, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  ALT, at Day 4 |  | 0.5 (2.43) | -0.8 (6.14)
  ALT, at Day 7 | 1.5 (2.83) | 0.5 (2.73) | 2.0 (7.91)
  ALT, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  ALT, at Day 8 |  | 0.8 (3.76) |
  ALT, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  ALT, at Day 10 |  | -1.0 (1.41) |
  ALT, at Day 14 | 1.0 (1.41) | 0.6 (2.13) | -2.0 (5.81)
  ALT, at Week 4 | 4.3 (6.34) | 1.6 (3.66) | -1.9 (8.18)
  ALT, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  ALT, at Week 16 | 4.4 (2.72) | 1.4 (2.45) | -0.1 (7.06)
  ALT, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  ALT, at Week 24 | 2.0 (4.44) | 1.3 (5.70) | -1.3 (5.96)
  AST, at Baseline | 14.5 (2.39) | 16.0 (2.98) | 18.1 (2.64)
  AST, at Day 2 | 0.4 (2.00) | 1.4 (1.77) | -1.8 (3.06)
  AST, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  AST, at Day 3 |  | 2.7 (1.63) | -0.6 (3.42)
  AST, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  AST, at Day 4 |  | 1.8 (1.72) | 0.5 (3.66)
  AST, at Day 7 | 2.8 (2.82) | 0.8 (3.06) | 2.5 (3.74)
  AST, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  AST, at Day 8 |  | 1.0 (3.03) |
  AST, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  AST, at Day 10 |  | -2.5 (0.71) |
  AST, at Day 14 | 1.9 (2.03) | 1.8 (2.76) | -0.9 (3.40)
  AST, at Week 4 | 3.0 (3.51) | 4.3 (8.96) | 0.0 (4.38)
  AST, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  AST, at Week 16 | 2.9 (1.81) | 1.1 (3.14) | 0.4 (3.95)
  AST, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  AST, at Week 24 | 2.0 (4.78) | 0.1 (2.47) | -0.7 (2.63)
  ALP, at Baseline | 54.6 (8.99) | 55.9 (20.00) | 57.1 (9.30)
  ALP, at Day 2 | 2.9 (3.83) | 0.6 (4.50) | -2.4 (4.44)
  ALP, at Day 3: number analyzed (Participants) | 0 | 6 | 8
  ALP, at Day 3 |  | 4.7 (4.03) | 0.0 (4.81)
  ALP, at Day 4: number analyzed (Participants) | 0 | 6 | 8
  ALP, at Day 4 |  | 4.0 (5.83) | 3.0 (3.89)
  ALP, at Day 7 | 4.6 (2.77) | 5.9 (4.05) | 4.9 (5.33)
  ALP, at Day 8: number analyzed (Participants) | 0 | 6 | 0
  ALP, at Day 8 |  | 6.8 (5.04) |
  ALP, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  ALP, at Day 10 |  | -1.5 (4.95) |
  ALP, at Day 14 | 7.6 (2.97) | 4.4 (4.17) | 2.8 (4.71)
  ALP, at Week 4 | 0.6 (6.50) | 7.9 (4.52) | -1.8 (2.76)
  ALP, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  ALP, at Week 16 | 4.8 (5.23) | 5.4 (5.42) | 1.0 (5.39)
  ALP, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  ALP, at Week 24 | -0.1 (5.17) | 3.3 (5.85) | 1.6 (4.89)

29. Secondary Outcome: Number of Participants With Worst Case Urinalysis at Post-baseline Compared With Baseline
Description: Urine samples were collected as assessed by protocol, at specific time points for laboratory analysis of VH3810109. At baseline and post-baseline, worst case urinalysis data was determined by comparing the resulted values of the urinalysis for each participant to the normal rage. This endpoint evaluates the changes from baseline for the worst case urinalysis.
Time Frame: Day 14 compared with baseline (Day -1)
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Participants
  Glucose | 1 | 0 | 0
  Protein | 0 | 1 | 1
  Leukocyte esterase | 0 | 1 | 1

30. Secondary Outcome: Change From Baseline in PR Interval, QRS Interval, QT Interval, and QT Interval Corrected for Heart Rate Using Fridericia's Formula (QTcF)
Description: ECG values were collected as assessed by protocol, at the indicated time points.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Miliseconds
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Miliseconds
  PR Interval, at Baseline | 161.375 (20.2762) | 164.000 (16.6733) | 164.875 (14.2872)
  PR Interval, at Day 1: number analyzed (Participants) | 8 | 0 | 8
  PR Interval, at Day 1 | -4.000 (10.7157) |  | 0.500 (4.5145)
  PR Interval, at Day 2 | -0.208 (7.5297) | 1.917 (9.5282) | 3.500 (7.6677)
  PR Interval, at Day 3 | 1.083 (7.8493) | 3.000 (10.6354) | 3.667 (10.6845)
  PR Interval, at Day 4 | 4.625 (8.6179) | 0.875 (10.8656) | 3.000 (10.0775)
  PR Interval, at Day 7 | 1.458 (11.6223) | 6.167 (10.9516) | 2.625 (6.3507)
  PR Interval, at Day 8: number analyzed (Participants) | 0 | 8 | 0
  PR Interval, at Day 8 |  | 5.875 (9.4330) |
  PR Interval, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  PR Interval, at Day 10 |  | 19.167 (8.7210) |
  PR Interval, at Week 4 | 9.542 (5.9038) | 4.250 (11.7700) | -2.250 (10.6231)
  PR Interval, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  PR Interval, at Week 24 | 4.583 (10.1164) | -0.958 (11.6571) | -1.905 (12.0872)
  QRS Interval, at Baseline | 92.875 (8.1141) | 90.750 (11.8291) | 100.250 (12.1155)
  QRS Interval, at Day 1: number analyzed (Participants) | 8 | 0 | 8
  QRS Interval, at Day 1 | 0.875 (3.5587) |  | -5.250 (6.8098)
  QRS Interval, at Day 2 | -2.292 (2.6693) | -0.458 (3.7116) | -3.708 (5.6833)
  QRS Interval, at Day 3 | -0.875 (2.3363) | -2.833 (6.2463) | -2.583 (3.6764)
  QRS Interval, at Day 4 | 1.458 (5.0895) | -1.875 (6.0708) | -4.458 (6.4855)
  QRS Interval, at Day 7 | 0.000 (5.1052) | -1.500 (6.8359) | -2.917 (6.3164)
  QRS Interval, at Day 8: number analyzed (Participants) | 0 | 8 | 0
  QRS Interval, at Day 8 |  | -1.042 (4.6987) |
  QRS Interval, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  QRS Interval, at Day 10 |  | -4.333 (6.5997) |
  QRS Interval, at Week 4 | 0.708 (3.9337) | -0.958 (3.8398) | -4.708 (6.2372)
  QRS Interval, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  QRS Interval, at Week 24 | -0.917 (4.5066) | -0.458 (4.4755) | -5.238 (6.4599)
  QT Interval, at Baseline | 378.875 (17.7719) | 395.875 (19.1493) | 380.375 (12.3513)
  QT Interval, at Day 1: number analyzed (Participants) | 8 | 0 | 8
  QT Interval, at Day 1 | 0.708 (12.1713) |  | -0.625 (8.6620)
  QT Interval, at Day 2 | 4.750 (12.1299) | 20.750 (18.9684) | 16.083 (13.6449)
  QT Interval, at Day 3 | 8.583 (18.2650) | 10.542 (27.0566) | 9.792 (12.7179)
  QT Interval, at Day 4 | 5.917 (22.1616) | 7.000 (27.0725) | 9.167 (18.5267)
  QT Interval, at Day 7 | 7.042 (20.7972) | 21.083 (21.4755) | 8.500 (13.6498)
  QT Interval, at Day 8: number analyzed (Participants) | 0 | 8 | 0
  QT Interval, at Day 8 |  | 19.167 (20.0206) |
  QT Interval, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  QT Interval, at Day 10 |  | 31.667 (55.1543) |
  QT Interval, at Week 4 | 14.083 (18.0614) | 31.167 (17.0023) | 10.583 (13.7318)
  QT Interval, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  QT Interval, at Week 24 | 15.125 (21.3348) | 13.167 (21.5318) | 15.952 (10.9771)
  QTcF Interval, at Baseline | 402.750 (10.5119) | 419.375 (13.7523) | 397.000 (14.8131)
  QTcF Interval, at Day 1: number analyzed (Participants) | 8 | 0 | 8
  QTcF Interval, at Day 1 | 2.833 (10.0570) |  | 1.375 (9.1780)
  QTcF Interval, at Day 2 | -1.875 (9.2923) | 1.083 (15.4486) | 3.375 (11.7924)
  QTcF Interval, at Day 3 | 0.917 (9.5232) | -1.250 (14.9047) | 2.083 (8.6295)
  QTcF Interval, at Day 4 | -2.000 (15.0449) | -4.292 (18.3220) | 1.917 (9.0847)
  QTcF Interval, at Day 7 | 8.667 (22.8341) | 0.958 (9.6715) | 3.500 (11.9004)
  QTcF Interval, at Day 8: number analyzed (Participants) | 0 | 8 | 0
  QTcF Interval, at Day 8 |  | 1.833 (14.8410) |
  QTcF Interval, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  QTcF Interval, at Day 10 |  | 0.667 (33.9411) |
  QTcF Interval, at Week 4 | 1.167 (10.6398) | 6.500 (8.8515) | 2.250 (8.4867)
  QTcF Interval, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  QTcF Interval, at Week 24 | 2.417 (10.5991) | 2.229 (14.8754) | 7.238 (5.6461)

31. Secondary Outcome: Change From Baseline in Temperature
Description: Temperature was measured at the indicated time points, in a supine position after the participant has been at rest for at least 5 minutes in a quiet setting without distractions.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Degrees Celcius
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Degrees Celcius
  Baseline | 36.54 (0.233) | 36.79 (0.344) | 36.49 (0.500)
  Day 2 | -0.10 (0.424) | -0.48 (0.437) | -0.14 (0.342)
  Day 3 | -0.23 (0.365) | -0.50 (0.475) | -0.25 (0.454)
  Day 4 | -0.03 (0.311) | -0.41 (0.569) | -0.20 (0.463)
  Day 7 | -0.05 (0.524) | -0.41 (0.622) | -0.04 (0.578)
  Day 8: number analyzed (Participants) | 0 | 8 | 0
  Day 8 |  | -0.41 (0.599) |
  Day 10: number analyzed (Participants) | 0 | 2 | 0
  Day 10 |  | -0.60 (0.566) |
  Day 14 | -0.13 (0.392) | -0.28 (0.492) | -0.28 (0.453)
  Day 21 | -0.11 (0.554) | -0.49 (0.352) | -0.04 (0.469)
  Week 4 | -0.21 (0.364) | -0.56 (0.534) | -0.09 (0.549)
  Week 8 | -0.28 (0.399) | -0.45 (0.535) | -0.20 (0.566)
  Week 12 | -0.23 (0.271) | -0.33 (0.607) | -0.28 (0.423)
  Week 16: number analyzed (Participants) | 8 | 8 | 7
  Week 16 | -0.34 (0.346) | -0.33 (0.575) | -0.69 (0.534)
  Week 20: number analyzed (Participants) | 7 | 8 | 7
  Week 20 | -0.17 (0.315) | -0.40 (0.414) | -0.19 (0.505)
  Week 24: number analyzed (Participants) | 8 | 8 | 7
  Week 24 | -0.19 (0.364) | -0.55 (0.678) | 0.09 (0.367)

32. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured at the indicated time points, in a supine position after the participant has been at rest for at least 5 minutes in a quiet setting without distractions.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Beats per minute (Beats/min)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Beats per minute (Beats/min)
  Baseline | 73.9 (7.85) | 71.1 (7.16) | 75.9 (12.26)
  Day 2 | -4.4 (6.74) | -7.6 (8.28) | -13.8 (10.66)
  Day 3 | -7.6 (4.84) | -5.4 (9.01) | -12.1 (8.63)
  Day 4 | -6.4 (7.76) | -4.3 (8.75) | -8.1 (11.52)
  Day 7 | -1.4 (18.68) | -9.4 (6.95) | -8.4 (14.81)
  Day 8: number analyzed (Participants) | 0 | 8 | 0
  Day 8 |  | -8.3 (5.78) |
  Day 10: number analyzed (Participants) | 0 | 2 | 0
  Day 10 |  | -12.0 (7.07) |
  Day 14 | -4.5 (7.60) | -10.0 (6.72) | -11.4 (16.95)
  Day 21 | -3.1 (11.43) | -9.1 (5.06) | -11.0 (18.45)
  Week 4 | -7.3 (3.28) | -9.9 (7.34) | -13.4 (12.05)
  Week 8 | -3.9 (15.13) | -8.0 (8.09) | -8.3 (15.75)
  Week 12 | -4.8 (10.44) | -6.3 (7.44) | -9.8 (14.21)
  Week 16: number analyzed (Participants) | 8 | 8 | 7
  Week 16 | -11.1 (10.25) | -5.1 (8.61) | -10.6 (10.66)
  Week 20: number analyzed (Participants) | 7 | 8 | 7
  Week 20 | -9.0 (8.14) | -5.0 (5.01) | -12.4 (8.06)
  Week 24: number analyzed (Participants) | 8 | 8 | 7
  Week 24 | -10.5 (6.57) | -4.3 (4.80) | -15.3 (11.50)

33. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Respiratory rate was measured at the indicated time points, in a supine position after the participant has been at rest for at least 5 minutes in a quiet setting without distractions.
Time Frame: From Baseline (Day -1) up to Week 24
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: Breaths per minute (Breaths/min)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Breaths per minute (Breaths/min)
  Baseline | 15.5 (1.41) | 15.8 (3.77) | 13.8 (1.98)
  Day 1/4 Hours Postdose: number analyzed (Participants) | 7 | 8 | 8
  Day 1/4 Hours Postdose | -1.4 (1.90) | -0.3 (3.45) | 2.0 (3.38)
  Day 1/8 Hours Postdose | 1.5 (2.56) | -2.3 (2.25) | 0.8 (3.85)
  Day 2 | -1.3 (3.20) | -2.0 (3.85) | 1.3 (2.12)
  Day 3 | -1.3 (2.12) | -1.5 (4.24) | 2.3 (2.71)
  Day 4 | -2.0 (2.14) | -1.5 (3.16) | 0.0 (2.62)
  Day 7 | 0.8 (4.77) | -2.8 (4.89) | -0.3 (2.92)
  Day 8: number analyzed (Participants) | 0 | 8 | 0
  Day 8 |  | -0.8 (5.01) |
  Day 10: number analyzed (Participants) | 0 | 2 | 0
  Day 10 |  | 0.0 (5.66) |
  Day 14 | -1.5 (2.98) | -2.0 (3.38) | -1.3 (2.12)
  Day 21 | -1.3 (2.60) | -2.3 (2.92) | 1.0 (3.85)
  Week 4 | 1.3 (2.38) | -2.0 (4.41) | 1.0 (2.83)
  Week 8 | 1.0 (2.83) | -2.3 (4.59) | 1.3 (1.83)
  Week 12 | -1.0 (2.14) | -2.5 (3.34) | 1.5 (2.33)
  Week 16: number analyzed (Participants) | 8 | 8 | 7
  Week 16 | -2.0 (4.28) | -2.5 (5.42) | 3.1 (1.95)
  Week 20: number analyzed (Participants) | 7 | 8 | 7
  Week 20 | -0.9 (3.80) | -1.0 (3.21) | 1.1 (3.98)
  Week 24: number analyzed (Participants) | 8 | 8 | 7
  Week 24 | -3.3 (2.38) | -2.5 (1.77) | 0.3 (2.93)

34. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Blood pressure was measured at the indicated time points, in a supine position after the participant has been at rest for at least 5 minutes in a quiet setting without distractions.
Time Frame: From Baseline (Day -1) up to Week 24
Population: Analysis was performed on PK set, who included participants who received study intervention and for whom valid and evaluable serum PK parameters were derived for the assesses timepoints and analysis.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
Number analyzed (Participants) | 8 | 8 | 8
Millimeters of mercury (mmHg)
  Systolic Blood Pressure, at Baseline | 112.8 (12.67) | 106.3 (11.68) | 114.4 (9.50)
  Systolic Blood Pressure, at Day 2 | -4.1 (12.24) | 3.5 (8.04) | -4.5 (7.19)
  Systolic Blood Pressure, at Day 3 | -2.9 (7.49) | 0.8 (5.99) | -4.5 (4.66)
  Systolic Blood Pressure, at Day 4 | -0.5 (9.20) | 0.3 (6.45) | -5.6 (6.23)
  Systolic Blood Pressure, at Day 7 | 2.1 (8.18) | 2.1 (6.03) | 3.6 (8.28)
  Systolic Blood Pressure, at Day 8: number analyzed (Participants) | 0 | 8 | 0
  Systolic Blood Pressure, at Day 8 |  | -2.4 (8.47) |
  Systolic Blood Pressure, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Systolic Blood Pressure, at Day 10 |  | 4.5 (13.44) |
  Systolic Blood Pressure, at Day 14 | 2.4 (8.68) | 11.3 (9.19) | 6.5 (10.38)
  Systolic Blood Pressure, at Day 21 | 5.4 (10.21) | 9.8 (13.36) | 7.8 (11.50)
  Systolic Blood Pressure, at Week 4 | -0.9 (8.54) | 9.5 (11.80) | 2.8 (7.85)
  Systolic Blood Pressure, at Week 8 | 9.0 (17.02) | 9.5 (14.43) | 5.6 (7.58)
  Systolic Blood Pressure, at Week 12 | -3.8 (4.89) | 4.5 (16.38) | 7.9 (11.54)
  Systolic Blood Pressure, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Systolic Blood Pressure, at Week 16 | 4.6 (5.55) | 7.9 (11.08) | -0.3 (10.27)
  Systolic Blood Pressure, at Week 20: number analyzed (Participants) | 7 | 8 | 7
  Systolic Blood Pressure, at Week 20 | -2.1 (14.28) | 2.1 (10.83) | 6.3 (7.83)
  Systolic Blood Pressure, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Systolic Blood Pressure, at Week 24 | 2.0 (7.78) | 6.4 (10.07) | -0.1 (4.91)
  Diastolic Blood Pressure, at Baseline | 66.5 (9.71) | 59.8 (6.45) | 62.1 (5.59)
  Diastolic Blood Pressure, at Day 2 | -1.6 (5.48) | 3.4 (8.23) | -0.5 (6.89)
  Diastolic Blood Pressure, at Day 3 | 2.4 (4.87) | 1.1 (7.24) | -1.9 (5.51)
  Diastolic Blood Pressure, at Day 4 | 0.6 (6.05) | -2.3 (4.62) | -0.8 (4.86)
  Diastolic Blood Pressure, at Day 7 | 1.9 (8.32) | -1.6 (4.41) | 9.5 (9.78)
  Diastolic Blood Pressure, at Day 8: number analyzed (Participants) | 0 | 8 | 0
  Diastolic Blood Pressure, at Day 8 |  | -1.8 (3.96) |
  Diastolic Blood Pressure, at Day 10: number analyzed (Participants) | 0 | 2 | 0
  Diastolic Blood Pressure, at Day 10 |  | 9.0 (8.49) |
  Diastolic Blood Pressure, at Day 14 | 1.6 (6.63) | 6.1 (3.72) | 6.1 (5.33)
  Diastolic Blood Pressure, at Day 21 | 2.8 (6.50) | 10.6 (8.37) | 12.9 (4.67)
  Diastolic Blood Pressure, at Week 4 | 2.1 (7.24) | 8.1 (6.40) | 7.6 (6.32)
  Diastolic Blood Pressure, at Week 8 | 6.4 (7.74) | 9.1 (3.44) | 7.6 (3.29)
  Diastolic Blood Pressure, at Week 12 | 0.5 (4.96) | 6.8 (7.15) | 11.5 (7.78)
  Diastolic Blood Pressure, at Week 16: number analyzed (Participants) | 8 | 8 | 7
  Diastolic Blood Pressure, at Week 16 | 3.8 (3.15) | 9.1 (5.11) | 8.4 (6.73)
  Diastolic Blood Pressure, at Week 20: number analyzed (Participants) | 7 | 8 | 7
  Diastolic Blood Pressure, at Week 20 | -2.0 (7.09) | 6.3 (5.55) | 13.6 (6.19)
  Diastolic Blood Pressure, at Week 24: number analyzed (Participants) | 8 | 8 | 7
  Diastolic Blood Pressure, at Week 24 | 1.5 (4.28) | 7.4 (6.57) | 12.1 (7.49)

ADVERSE EVENTS:
Time Frame: SAEs, all cause mortality and non-SAEs were collected from Day 1 post-administration up to Week 24.
Arm/Group | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] | Part 2 Group: VH3810109 60 mg/kg [IV] | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC]
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 8/8 | 1/8 | 8/8
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Group: VH3810109 20 mg/kg + rHuPH20 [SC] (N=8) | Part 2 Group: VH3810109 60 mg/kg [IV] (N=8) | Part 3 Group: VH3810109 3000 mg + rHuPH20 [SC] (N=8)
Injection site erythema (General disorders) | 7 (7) | 0 (0) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 1 (1) | 0 (0) | 2 (2)
Injection site pruritus (General disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Medical device site dermatitis (General disorders) | 0 (0) | 1 (1) | 0 (0)
Injection site bruising (General disorders) | 0 (0) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site induration (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT05291520/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/20/NCT05291520/SAP_001.pdf